CLINICAL TRIAL: NCT03962283
Title: Rifaximin and Misoprostol Combination Therapy for Healing of Small Bowel Ulcers in Aspirin Users With Small Bowel Bleeding: A Double Blind Randomized Trial
Brief Title: Rifaximin and Misoprostol Combination Therapy for Healing of Small Bowel Ulcers in Aspirin Users
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MISO RF
Record Dates: First submitted 2019-05-19; First posted 2019-05-24 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Small Bowel Disease; Rifaximin
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rifaximin (Active Comparator): ASA daily + misoprostol + Rifaximin (Rifaximin group)
  Interventions: Drug: Rifaximin
- Rifaximin Placebo (Placebo Comparator): ASA daily + misoprostol + Placebo Rifaximin (Placebo group)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 200mcg four times daily
  Arms: Rifaximin
Drug: Placebo oral tablet — Placebo Rifaximin four times daily
  Arms: Rifaximin Placebo

SUMMARY:
Background: Investigators have previously shown that misoprostol can heal small bowel ulcers in aspirin users with small bowel bleeding. However, the rate of small-bowel mucosal healing was low with use of misoprostol alone. There is evidence to suggest that bacteria contribute to the development aspirin-induced ulcers and antibiotics may be useful in its treatment. Rifaximin, a non-absorbed oral antibiotic that target the gastrointestinal tract have been shown to be safe and effective in a few other gastrointestinal conditions.

Small bowel capsule is the most sensitive and non-invasive way to investigate the small bowel. It plays an important role in obscure GIB investigations.

Aims: The aim of this randomized study is to test the hypothesis that misoprostol combined with rifaximin is superior to misoprostol alone for healing of small bowel ulcers in aspirin users complicated by small bowel bleeding.

Study design: 8-week double-blind randomized trial

DETAILED DESCRIPTION:
Aspirin is one of the most commonly prescribed drugs worldwide It is widely used as the first line agent for prevention and treatment of heart diseases and stroke. It is well recognized that aspirin and other non-steroidal anti-inflammatory drugs (NSAIDs) are associated with risk of upper gastrointestinal (the stomach) bleeding. It is increasingly recognized to have adverse effects in the small bowel, including ulcers resulting in bleeding.

Bleeding from the small bowel has been very difficult to diagnose as it is beyond the reach of the conventional endoscopy. But with advances in endoscopic technique, video capsule endoscopy is now available to visualize the whole of the digestive tract. Capsule endoscopy is the size and shape of a pill which contains a tiny camera. After ingesting the capsule, pictures are taken inside of the gastrointestinal tract. Capsule endoscopy is now recommended to be a noninvasive test to identify source of small bowel bleeding.

Investigators have recently shown that misoprostol can heal small bowel ulcers in aspirin users with small bowel bleeding. However, the complete healing rate with misoprostol alone was only 40%. This suggests that we should continue to investigate for additional therapies in order to achieve higher success rate of healing of aspirin-induced small bowel ulcers.

Rifaximin is a non-absorbed oral antibiotic that targets the gastrointestinal tract. It was first described in 1982 and introduced into the Italian market 5 years later. Since then, rifaximin has had U.S. Food and Drug Administration (FDA) approval for treatment of travellers' diarrhea (year approved = 2004), hepatic encephalopathy (year approved=2010), irritable bowel syndrome (IBS) with diarrhea (year approved= 2015). Unlike the systematically available antibiotics, it allows localized enteric targeting of pathogens and is associated with minimal risk of systemic toxicity or side effects. In addition, the restricted use of non-absorbed oral antibiotics should also reduce the development of wide spread resistance.

The aim of this study is to test the hypothesis that the combination therapy of rifaximin and misoprostol is superior to misoprostol alone for healing of small bowel ulcers in aspirin users complicated by small bowel bleeding.

Participants are invited to this study because some predefined lesions are detected by the small bowel capsule endoscopy. Participants will be randomly assigned to receive either a combination therapy of misoprostol and rifaximin or misoprostol and rifaximin placebo for 8 weeks. Participants will be contacted by telephone after 1 week for any adverse events. Participants will then return at Week 8 to undergo a follow-up capsule endoscopy. Lab tests, drug compliance, and adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Suspected small bowel overt bleeding - melena or hematochezia with or without a source of bleeding from gastroscopy and colonoscopy or suspected small bowel occult blood loss - defined as a significant decrease in hemoglobin (> 2g/dL), without a source of bleeding from gastroscopy and colonoscopy, confirmed iron deficiency anemia, and absence of other identifiable causes for hemoglobin decrease (e.g. fluid overload, progressive renal failure, malnutrition, or other hematological disorders such as hemolysis or malignancies)
* Continuous use of aspirin for the duration of the trial
* Age ≥ 18
* Written informed consent obtained

Exclusion Criteria:

* Increased risk of capsule retention (e.g. gastric outlet obstruction, bypass surgery, Crohn's disease or suspected small bowel stricture)
* Abnormal findings on gastroscopy that may account for bleeding episode: clean-based ulcer >2 cm or >5 erosions, esophageal varices, grade C or D erosive esophagitis, vascular malformations
* Unable to swallow the capsule endoscopy
* Terminal illness
* Concomitant use of NSAIDs, sucralfate, rebamepide, antibiotics, corticosteroids (prednisolone >7.5 mg daily or equivalent), and iron supplement
* Pregnancy (except LMP within 7 days) or women of child-bearing age without regular use of contraception
* Contraindications to colonoscopy or capsule endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Healing of small bowel ulcers | 8 weeks after randomization
  Capsule endoscopy will be performed to check if there is complete healing of small bowel ulcers, with or without red spots.

SECONDARY OUTCOMES:
Change in numbers of ulcer/erosions | 8 weeks after randomization
  Change in numbers of ulcer/erosions from baseline within and between groups
Change in blood hemoglobin level | 8 weeks after randomization
  Change in blood hemoglobin level from baseline within and between groups

CONTACTS AND LOCATIONS:
Overall Officials: Francis Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China
- Prince of Wales Hospital, Hong Kong, Hong Kong